CLINICAL TRIAL: NCT03922412
Title: Plantar Compartment Block Versus Sciatic Block in Hallux Valgus Ambulatory Surgery : a Prospective, Randomised, Double Blind Study
Brief Title: Plantar Compartment Block Versus Sciatic Block in Hallux Valgus Ambulatory Surgery
Acronym: Plantar-block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RECHMPL18_0489
Record Dates: First submitted 2019-04-11; First posted 2019-04-22 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia
Keywords: Anesthesia; plantar Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plantar block (Active Comparator): Short lasting sciatic nerve block (mepivacaine 1% 200mg) and long lasting plantar block (ropivacaine 0,5% 25mg + 2mg dexamethasone) with distal deep peroneal block (ropivacaine 0,5% 2ml).
  Interventions: Procedure: PLANTAR BLOCK
- Sciatic popliteal block (Active Comparator): Long lasting sciatic nerve block (ropivacaine 0,5% 100mg + 2mg dexamethasone)
  Interventions: Procedure: Sciatic popliteal block

INTERVENTIONS:
Procedure: PLANTAR BLOCK — 1. Sciatic popliteal block : patient in lateral position, injection of 20 ml of the mixture labelled " BLOC POPLITE " containing 20 ml of mepivacain 1% (200mg)
  2. Plantar block 10 minutes later : patient in supine position. Medial midfoot injection of 5 ml of the mixture labelled " BLOC PLANTAIRE " containing 5 ml of Ropivacaine 0,5% (25mg) with 0,5 ml dexaméthasone (2mg)
  3. Distal deep fibular block : patient in supine position, injection around the dorsal foot artery of 2 ml of the mixture labelled " BLOC FIBULAIRE " containing 2 ml of Ropivacaine 0,5% (10mg).
  Arms: plantar block
Procedure: Sciatic popliteal block — 1-Sciatic popliteal block : patient in lateral position, injection of 20 ml of the mixture labelled " BLOC POPLITE " containing 20 ml of ropivacaine 0,5% (100mg) with 2mg (0,5 ml) of dexamethasone
  Arms: Sciatic popliteal block

SUMMARY:
Hallux valgus surgery is known as a painful surgery. Qualitative pain management is the key to successful early recovery and rehabilitation.

Sciatic popliteal nerve block is widely used despite the risk of falling due to prolonged motor blockade.

Plantar block combined with distal peroneal block may be a better analgesic option in order to provide fast track rehabilitation.

This study aims to determine the quality of deambulation following hallux valgus surgery.

Block quality, post operative pain, patient satisfaction and length of hospital stay will be compared in this study.

Patients scheduled for ambulatory (hallux valgus) surgery under regional anaesthesia alone (without general anesthesia) will be recruited.

Consenting patients will be randomized the day of surgery to one of those two groups :

1. Short lasting sciatic nerve block (mepivacaine 1% 200mg) and long lasting plantar block (ropivacaine 0,5% 25mg + 2mg dexamethasone) with distal deep peroneal block (ropivacaine 0,5% 2ml).
2. Long lasting sciatic nerve block (ropivacaine 0,5% 100mg + 2mg dexamethasone)

All patients will benefit from post operative analgesia including paracetamol, nonsteroidal antiinflammatory drugs intravenously.

During PACU stay, pain will be assessed using the VAS (visual analogue scale) score, and analgesic IV consumption.

Temporospatial gait analysis will be assessed with a GAITRITE system before the patient leave the hospital.

Deambulation and walking ability will be evaluated at home postoperatively to day 3 using an acetimetry bracelet.

Pain, postoperative analgesic requirement, sleep quality and overall patient satisfaction (EVAN-LR) will also be assessed during the first 3 postoperative days.

DETAILED DESCRIPTION:
Hallux valgus surgery is known as a painful surgery. Qualitative pain management is the key to successful early recovery and rehabilitation.

Sciatic popliteal nerve block is widely used despite the risk of falling due to prolonged motor blockade.

Plantar block combined with distal peroneal block may be a better analgesic option in order to provide fast track rehabilitation.

This study aims to determine the quality of deambulation following hallux valgus surgery.

Block quality, post operative pain, patient satisfaction and length of hospital stay will be compared in this study.

Patients scheduled for ambulatory (hallux valgus) surgery under regional anaesthesia alone (without general anesthesia) will be recruited.

Consenting patients will be randomized the day of surgery to one of those two groups :

1. Short lasting sciatic nerve block (mepivacaine 1% 200mg) and long lasting plantar block (ropivacaine 0,5% 25mg + 2mg dexamethasone) with distal deep peroneal block (ropivacaine 0,5% 2ml).
2. Long lasting sciatic nerve block (ropivacaine 0,5% 100mg + 2mg dexamethasone)

All patients will benefit from post operative analgesia including paracetamol, nonsteroidal antiinflammatory drugs intravenously.

During PACU stay, pain will be assessed using the VAS (visual analogue scale) score, and analgesic IV consumption.

Temporospatial gait analysis will be assessed with a GAITRITE system before the patient leave the hospital (6 hours after ALR).

Deambulation and walking ability will be evaluated at home postoperatively to day 3 using an acetimetry bracelet.

Pain, postoperative analgesic requirement, sleep quality and overall patient satisfaction (EVAN-LR) will also be assessed during the first 3 postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* patient covered by social health insurance
* have signed written informed consent
* scheduled for hallux valgus ambulatory surgery

Exclusion Criteria:

* protected patients or patients incapable of giving written informed consent
* pregnant or breastfeeding woman
* vulnerable adult
* inability to participate in pain scoring scales
* severe coagulopathy
* allergy or contraindications to study drugs
* preoperative gait disorders
* chronic kidney disease with glomerular filtration rate (GFR) ≤ 50 ml/min (estimated by the Cockcroft and Gault formula)
* severe chronic liver disease
* chronic pain (treated by non steroidal anti inflammatory drugs, opioids, neuroleptic drugs, antidepressant or anticonvulsants)
* peripheral neuropathy
* intervention under general anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
Number of steps walking ability assessed by GAITRITE Test | 6 hours after ALR
  Comparison of the deambulation assessed by GAITRITE test (walking test) between patient who received plantar block and patient who received sciatic popliteal block

SECONDARY OUTCOMES:
Quantity of postoperative rescue analgesics taken | up to 3 days after surgery
  Comparison of the postoperative pain assessed by the Quantity of post-operative rescue analgesics between each group of patients
Assessment of the quality of the sensory blocks | during the surgery
  Comparison of the sensory territories of anesthesia using cold between each group
Assessment of the patient hospitalisation duration | up to 3 days after surgery
  Comparison of the duration of hospitalization between each group
Assessment of overall patient satisfaction assessed by the scale EVAN Loco regional | up to 3 days after surgery
  Comparison of overall patient satisfaction between each group
Assessment of sleep quality Assessment of patient sleep quality | up to 3 days after surgery
  Comparison of patient sleep quality assessed by the somnifer consumption during the postoperative hospitalization between each group
Efficacity of patient walking ability | up to 3 days after surgery
  Comparison of the deambulation assessed by acetemeter between patient who received plantar block and patient who received sciatic popliteal block

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided